CLINICAL TRIAL: NCT04555967
Title: SAPIEN 3 Ultra System Post-Market Clinical Follow-up Study
Brief Title: SAPIEN 3 Ultra System PMCF
Status: Active, not recruiting | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-09
Record Dates: First submitted 2020-09-01; First posted 2020-09-21 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Aortic Valve Stenosis
Keywords: Transcatheter Aortic Valve Implantation; Transcatheter Aortic Valve Replacement; SAPIEN 3 Ultra
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Transcatheter aortic valve implantation
  Interventions: Device: SAPIEN 3 Ultra System

INTERVENTIONS:
Device: SAPIEN 3 Ultra System — Transcatheter aortic valve implantation

SUMMARY:
A post-market study of the Edwards SAPIEN 3 Ultra System in subjects with symptomatic, severe, calcific aortic stenosis.

DETAILED DESCRIPTION:
To monitor and review device performance and outcomes of the SAPIEN 3 Ultra System in subjects with symptomatic, severe, calcific aortic stenosis.

ELIGIBILITY:
1. Subject meets the criteria per the Indication and Contraindications according to the current IFUs.

   * Indication for Use: The Edwards SAPIEN 3 Ultra THV, the Edwards SAPIEN 3 THV, and the associated delivery systems are indicated for use in patients with severe, symptomatic, calcific aortic valve stenosis who are judged by a Heart Team, to be at intermediate or greater risk for open surgical therapy (i.e., predicted risk of surgical mortality ≥ 3% at 30 days, based on the STS risk score and other clinical comorbidities unmeasured by the STS risk calculator).
   * Contraindications: Evidence of intracardiac mass, thrombus, vegetation, active infection or endocarditis; Inability to tolerate anticoagulation/antiplatelet therapy.
2. Subject has provided written informed consent to comply with all study procedures and follow-up visits

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with symptomatic, severe, calcific aortic stenosis treated per the indications for use in the Instructions for Use
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Device success per VARC-3, defined as meeting all of the following: | 30 days
  * Technical success
  * Freedom from mortality
  * Freedom from surgery or intervention related to the device or to a major vascular or access-related, or cardiac structural complication
  * Intended performance of the valve (mean gradient < 20 mmHg, peak velocity < 3 m/s, Doppler velocity index ≥ 0.25, and less than moderate aortic regurgitation)

SECONDARY OUTCOMES:
Death | 1 year
Stroke | 30 days and 1 year
Major vascular complications | 30 days
Life threatening bleeding | 30 days
New conduction defects requiring permanent pacemaker | 30 days
Acute kidney injury stage 2-3 | 7 days
New onset atrial fibrillation | 30 days
Rehospitalization (valve-related or due to worsening heart failure) | 1 year
Paravalvular leak | 30 days and 1 year
Mean aortic valve gradient | 30 days and 1 year

CONTACTS AND LOCATIONS:
Locations (11):
- Medizinische Universitaet Wien, Vienna, Austria
- St. Paul's Hospital Vancouver, Vancouver, British Columbia, Canada
- Aarhus University Hospital, Skejby, Aarhus, Denmark
- Helsinki University Hospital, Helsinki, Finland
- Germany (3):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Deutsches Herzzentrum Berlin, Berlin
  - Universitares Herzzentrum Hamburg, Hamburg
- Ospedale G. Pasquinucci, Massa, Italy
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- United Kingdom (2):
  - Royal Victoria Hospital Belfast, Belfast
  - King's College Hospital London, London

IPD SHARING:
Plan to Share IPD: No